CLINICAL TRIAL: NCT07259369
Title: The Effects of an App-based Acupressure Intervention on Alleviating Fatigue, Pruritus, and Sleep Quality Among Hemodialysis Patients
Brief Title: The Effects of an App-based Acupressure on Alleviating Fatigue, Pruritus, and Sleep Quality Among Hemodialysis Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University (Other)
Responsible Party: Principal Investigator, NGUYEN THI THUY NGA, PhD student, Taipei Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 025-462/DD-YTCC
Record Dates: First submitted 2025-11-17; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Hemodialysis Patient; Fatigue
Keywords: chronic kidney disease; fatigue; App; pruritus; self-acupressure; sleep quality
MeSH Terms: conditions — Fatigue; Renal Insufficiency, Chronic; Alzheimer Disease; Pruritus; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- App-based acupressure Group (Experimental): The intervention group will use an app-based self-guided acupressure program to do the acupressure by themselves once daily for 4 weeks.
  Interventions: Device: app-based acupressure
- Control group (No Intervention): Participants in the control group will receive usual care and no other intervention. After completing the 12-week study, they will be granted free access to the application.

INTERVENTIONS:
Device: app-based acupressure — The intervention group will use an app-based self-guided acupressure program to do the acupressure by themselves once daily for 4 weeks. The app is structured into two main modules: Introduction and Practice. The Introduction section provides basic information about acupressure, including its definition, health benefits, and important safety considerations. This content is delivered through text, photos, and video to support different learning preferences.
  Arms: App-based acupressure Group

SUMMARY:
Objectives: To evaluate the effectiveness of an app-based self-guided acupressure intervention in alleviating fatigue and pruritus, and in improving sleep quality among hemodialysis patients.

Design and subjects: The parallel randomized controlled trial will be employed in one hospital. Block randomization in a 1:1 ratio will be used to assign the patients to the intervention and control groups. It is estimated that 50 to 100 participants receiving hemodialysis will be recruited.

Instrument: The demographic and health-related information questionnaire, the Post-dialysis Fatigue (PDF), 5-D Itch, and Pittsburgh Sleep Quality Index will be used in this study.

Interventions: The intervention group will use an app-based self-guided acupressure program to do the acupressure by themselves once daily for 4 weeks. Participants in the control group will receive usual care and no other intervention.

Data analysis: Both intention-to-treat and per-protocol analysis approaches will be performed. Generalized Estimating Equations (GEE) analysis will be used to assess the effectiveness of the interventions. Sensitivity analysis will be conducted to assess the impact of missing data on the treatment effect if necessary.

Expected outcomes: Participants in the intervention group will know how to do the self-guided acupressure by themselves. If the intervention is effective, the App can be introduced to the hemodialysis patients who need it.

DETAILED DESCRIPTION:
Introduction Fatigue is a multidimensional construct, encompassing behavioral, emotional, sensory, and cognitive domains (Joshwa et al., 2020). Among patients receiving hemodialysis (HD), fatigue is one of the most commonly reported and debilitating symptoms (Bossola et al., 2023). This symptom profoundly affects patients' functional capacity, psychological well-being, and overall quality of life (Bossola et al., 2023).

The effectiveness of both pharmacological and non-pharmacological interventions for managing fatigue in hemodialysis patients remains inconsistent due to a lack of high-quality evidence (Natale et al., 2023). Pharmacological options, such as erythropoiesis-stimulating agents, serotonin reuptake inhibitors, beta-blockers, anabolic steroids, and glucose-enriched dialysate, have produced mixed results (Natale et al., 2023). Similarly, non-pharmacological approaches, including amino acid supplementation, music therapy, meditation, cognitive-behavioral therapy, exercise, nutritional support, and light therapy, have shown limited and inconclusive benefits (Natale et al., 2023). Other interventions, such as increasing the frequency of dialysis sessions, adjusting blood flow rates, and home blood pressure monitoring, have also been explored, but lack strong supporting evidence (Natale et al., 2023). Given the complex nature of fatigue in this population, further well-designed studies and interventions are needed to establish effective management strategies.

Acupressure, a non-invasive technique derived from traditional Chinese medicine, has been explored as a potential non-pharmacological approach for reducing fatigue across various domains, such as behavioral, emotional, sensory, and cognitive fatigue (Chang et al., 2024). Acupressure can be performed by patients themselves after appropriate training, rather than relying on a therapist. Self-administered acupressure is time-efficient, low-cost, and easy to learn. Several studies have investigated its use for managing insomnia disorder (Yeung et al., 2022), pain in patients with osteoarthritis (Guo et al., 2021; Yeung et al., 2024), cancer-related fatigue in breast cancer survivors (Zick et al., 2016), quality of life in patients with perennial allergic rhinitis (Li et al., 2023), and anxiety levels in prediabetic women (Haghighat et al., 2024). Recently, a pilot RCT demonstrated that self-acupressure is safe and feasible for preventing respiratory tract infections in patients with chronic kidney disease (CKD) (Liu et al., 2022) and for managing symptoms and improving quality of life in HD patients (Parker et al., 2024).

The rapid advancement of mobile health (mHealth) technologies has significantly enhanced both the accessibility and personalization of healthcare. Smartphone applications, in particular, have become valuable tools for promoting self-care and managing chronic conditions (Sockolow et al., 2021; Wang et al., 2021) through features such as personalized goal setting, timely reminders, social interaction, and supportive feedback (Yi et al., 2018). A systematic review indicated that app-based mHealth interventions can effectively reduce stress and enhance self-management among non-clinical and subclinical populations (Sîrbu & David, 2024). Moreover, app-based interventions demonstrate their superiority in reducing fatigue among HD patients. A previous randomized controlled trial demonstrated that a recreational therapy app significantly reduced fatigue levels compared to standard care (Alishahi et al., 2024). The app provided a variety of content, including music, comedy, exercise, and educational materials, to help patients manage various dimensions of fatigue.

Although previous studies have shown that acupressure can effectively reduce fatigue, most studies have relied on trained therapists to administer the treatment. This limits accessibility and long-term sustainability, particularly for those who need ongoing symptom management. Although growing interest in digital health solutions, few studies have explored the use of mobile applications to guide self-administered acupressure as a convenient, cost-effective, and scalable alternative. App-based platforms can empower patients by enabling consistent practice and offering immediate, guided instruction without the need for direct clinical supervision. This approach, combining traditional therapies with modern digital tools, may enhance patient self-management and improve fatigue-related outcomes. Therefore, the primary aim of this study is to evaluate the effectiveness of an app-based self-guided acupressure intervention in alleviating fatigue among patients undergoing hemodialysis. The secondary aims are to examine its effects on pruritus and sleep quality in the same population. The hypotheses of this study are:

H1: Hemodialysis patients who receive the app-based self-guided acupressure will have greater fatigue relief compared to those receiving usual care.

H2: Hemodialysis patients who receive the app-based self-guided acupressure will have greater pruritus relief compared to those receiving usual care.

H3: Hemodialysis patients who receive the app-based self-guided acupressure will have greater improvement in sleep quality compared to those receiving usual care.

2. Theoretical approach Bandura's Social Cognitive Theory, with a central focus on the construct of self-efficacy (Bandura, A., 1977), will be used to develop the self-guided acupressure apps (Figure 1). Self-efficacy theory explains how individuals develop and modify beliefs in their ability to perform specific behaviors, and how these beliefs influence behavioral change, performance outcomes, and personal well-being. According to Bandura, expectations of personal efficacy are derived from four principal sources of information: performance accomplishments, vicarious experience, verbal persuasion, and physiological and emotional states (Bandura A., 1977). The self-acupressure app in this study is intentionally designed to address each of these four domains: The app encourages users to engage in regular, structured self-acupressure sessions. As participants complete these sessions, they experience successive mastery, which reinforces their confidence in managing fatigue through their own actions. Second, the app includes guided video demonstrations of self-acupressure techniques, allowing participants to observe others performing the same tasks. This modeling helps cultivate the belief that "if others can do it, so can I." Third, the app integrates motivational pop-up messages, such as "Well done!" or "Almost there-don't give up now!", to encourage continued engagement and reinforce users' belief in their ability to succeed, particularly during moments of low motivation. Finally, as acupressure helps reduce physical fatigue and promotes relaxation, users experience positive internal states. These improvements contribute to more favorable self-efficacy judgments and further motivate sustained engagement in self-care behaviors. By enhancing users' self-efficacy, the app aims to increase confidence in managing fatigue and foster long-term self-management among patients receiving hemodialysis.

Study design This study is a two-arm parallel randomized controlled trial (RCT). The CONSORT (Consolidated Standards of Reporting Trials) guidelines will be used to report this study. This study will be prospectively registered at ClinicalTrials.gov (https://clinicaltrials.gov/) prior to participant enrollment.

3.2 Research setting and participants The study will be conducted in the hemodialysis unit in Hoe Nhai Hospital, Hanoi, Vietnam. The patients are 18 years old or over, are able to speak and understand Vietnamese, receive hemodialysis at least three times a week for three months or longer, have a score equal to or greater than 4 on a numeric rating scale (NRS, 0-10) (Oldenmenger et al., 2013), has a smartphone or tablet, and can provide written informed consent. The patients who have advanced cancer, cognitive impairment, chronic obstructive pulmonary disease, severe edema, have already used or plan to use acupressure or acupuncture in the following 3 months, or have soft tissue or vascular disease in their lower extremities will be excluded.

Sample size will be calculated using G*Power software version 3.1.2 (Faul et al., 2009). With a power of 0.80, a 2-sided significance level of 5%, and a medium effect size of 0.35 (Vagharseyyedin et al., 2019), it was estimated that a total sample size of 42 participants would be needed. In addition, the attrition rate of 20% will be considered. Finally, we will recruit 50 to 100 participants in this study.

3.3 Instruments The questionnaires include demographic and health-related information, Post-Dialysis Fatigue Scale, 5-D Itch, Pittsburgh Sleep Quality Index, and Hemodialysis Comfort Scale version II.

3.3.1 Demographic and health-related information questionnaire This questionnaire consists of gender, age, employment status, marital status, educational level, economic status, duration of dialysis, comorbidities, self-assessed health status, exercise frequency, BMI, Kt/V, serum phosphorus, serum potassium, serum albumin, interdialytic gain weight (IDGW), blood pressure before and after dialysis (to calculate intradialytic hypertension). The self-assessed health status was measured on a five-point scale from 1 to 5 (1 = poor, 2 = fair, 3 = good, 4 = very good, 5 = excellent). These variables will be used to analyze the differences between the two groups at the baseline.

3.3.2 Post-Dialysis Fatigue scale (PDF) PDF, developed by Hirotoshi Kodama et al. (2020), will be used to measure fatigue in this study. This scale comprises 13 self-reported items rated on a five-point Likert scale, ranging from 1 (strongly agree) to 5 (not at all). The score will be reversed for analysis, and the total score is between 13 and 65, with higher scores indicating more severe fatigue. The PDF scale is concise and can be completed in 5-10 minutes. The Vietnamese version questionnaire translated by the researchers will be used in this study. Its content validity index (CVI) is 0.99, and Cronbach's alpha is 0.90.

3.3.3 5-D Itch The 5-D Itch was developed by Elman et al. (2010) to evaluate the severity of skin itching conditions over the past 2 weeks based on five dimensions: duration, degree, direction, disability, and distribution. Itching at up to two sites receives a score of 1; three to five sites are assigned a score of 2; the score is 3 for six to ten sites; 11 to 13 sites are scored 4; and the highest score of 5 is given for 14 to 16 sites. The total scores range from 5 to 25. Higher scores indicate greater itch severity. The scale of the Vietnamese version demonstrated good content validity (CVI=1.00) and acceptable reliability with Cronbach's α of 0.80.

3.3.4 Pittsburgh Sleep Quality Index (PSQI) The PSQI was developed by Buysse et al. (1989) consists of 7 components, 3 factors, and 19 subitems, and aims to evaluate a person's sleep quality within the last month, including seven components: (1) subjective sleep quality, (2) sleep latency, (3) sleep duration, (4) habitual sleep efficiency, (5) sleep disturbances, (6) use of sleeping medication and (7) daytime dysfunction. Component scores range from 0 (no difficulty) to 3 (severe difficulty). The total score ranges from 0 to 21, with higher values indicating poor sleep quality. A score of more than 5 indicated a person had poor quality sleep. The Vietnamese version will be used in this study and has a Cronbach's alpha coefficient of 0.789, indicating an acceptable internal consistency (To, 2017).

3.4 Intervention 3.4.1 Intervention group Participants in the intervention group will be instructed to download and install the mobile application, with initial training provided by the research team to ensure correct usage. During the training session, participants will be guided through the app's features, including how to navigate the interface, initiate acupoint stimulation, respond to reminder notifications, and record daily activity logs. Participants will also be asked to perform a return demonstration using the app and will have the opportunity to ask questions to clarify any uncertainties. Ongoing support will be provided throughout the study via Zalo, allowing participants to contact the RA if they have any problems with the app.

The app will send scheduled pop-up notifications twice each evening (within a 10-minute interval) to remind participants to perform acupressure as instructed in the app. Participants will be required to record the number of stimulations completed per session directly within the app.

Compliance will be monitored through the app's internal logging system, which tracks user-reported activity in real time. If a participant fails to meet the minimum daily requirement (one session per day, each consisting of one minute of stimulation per acupoint), the system will trigger additional reminder notifications. The application also employs a motivational feedback mechanism: participants with high adherence (≥80% of prescribed sessions) will receive positive reinforcement messages such as "Well done!" while those with lower adherence (<80% or no practice within 3 consecutive days) will receive motivational prompts such as "Almost there. Don't give up now!" to promote ongoing involvement.

3.4.1.1 Acupoints selection The self-administered acupressure includes four acupoints, namely, Sanyinjiao (SP6), Yongquan (KI1), and Zusanli (ST36), Yin Tang (GV29) acupoints selected based on the previous systematic reviews (Chang et al., 2024; Hsieh et al., 2023; Vagharseyyedin et al., 2019) and the theoretical basis of traditional Chinese medicine (Zhang et al., 2014). The location of each acupoint is shown in the table below (Table 1) (Liang, 2016; WHO, 2008).

Table 1. Location of acupoints No Acupoints Location

1. Sanyinjiao (SP6) (Tam Âm Giao) On the tibial aspect of the leg, posterior to the medial border of the tibia, 3 B-cun superior to the prominence of the medial malleolus.

   Note: 1 B-cun superior to KI8.
2. Yongquan (KI1) (Dũng Tuyền) On the sole of the foot, in the deepest depression of the sole when the toes are ﬂexed. Note: When the toes are ﬂexed, KI1 is located approximately in the depression at the junction of the anterior one-third and the posterior two-thirds of the line connecting the heel with the web margin between the bases of the second and third toes.
3. Zusanli (ST36) (Túc Tam Lý) On the anterior aspect of the leg, on the line connecting ST35 with ST41, 3 B-cun inferior to ST35.

   Note: ST36 is located on the tibialis anterior muscle.
4. Yin Tang (GV29) (Ấn đường) At the center of the glabella, on the anterior midline, between the eyebrows.

3.4.1.2 Operation of acupressure Participants will be asked to engage with the app once daily at a time that is convenient for them, preferably before going to bed. During each session, they will view the app and follow the instructions provided by the app to stimulate designated acupoints for a duration of one minute per acupoint. Each acupoint will be stimulated bilaterally, applying 2 rotations by finger or equipment per second. As a result, each session will involve a total of 7 acupoints with 7 minutes of stimulation. The total intervention period will span four weeks.

3.4.1.3 Developing an app-based self-guided acupressure intervention (AcuCare) 3.4.1.3.1 Interface of the application The app is structured into two main modules: Introduction and Practice. The Introduction section provides basic information about acupressure, including its definition, health benefits, and important safety considerations. This content is delivered through text and video to support different learning preferences.

The Practice section focuses on hands-on guidance, covering four commonly used acupressure points. Each point is represented as a selectable item, leading to a detailed view that includes: (1) an image showing the exact location of the point; (2) an introductory instructional video; and (3) a written transcript of the video content for users who prefer to read. Additionally, a prominent action button on this screen allows users to access a second, more detailed video. This second video is designed to guide the user through the practice step-by-step, in real time, making it easier to follow along and apply the technique correctly.

Self-Acupressure Instruction Procedure

1. Preparation:

   * Comfort room, a bed/chair
   * Shorten fingers' nails
   * Acupressure tools (if needed)
2. Implementation

   * Hand washing
   * Posture: sitting position on a bed/chair.
   * Identify the acupoint location
   * Pressing and applying 2 rotations by finger or equipment per second until you feel "de qi". Applying for 1 min at each acupoint.
3. Monitoring And Managing Complications Gently massage the painful area, reducing the impact on the treatment area. The procedure may be stopped if the body is too sensitive to the effects.

   3.4.1.3.2 Fidelity of self-guided acupressure training App All the program content will be reviewed and approved by the 2 experts who are registered Chinese medicine doctors and 3 nephrologists with at least 5 years' clinical experience and at least a Master's degree.

   3.4.2 Control group Participants assigned to the usual care group will receive the standard care routinely provided for their condition. They will not engage with the study-specific mobile application or any experimental procedures. However, after completing the 12-week study, they will be granted free access to the application.
4. Data collection 4.1 Data collection procedure Participants will be randomly assigned to study groups using block randomization to ensure balanced allocation across groups. A research assistant, who is not involved in participant recruitment, data collection, or analysis, will generate the random allocation sequence using a computer-based randomization tool. To maintain allocation concealment, the assignments will be placed in consecutively numbered, sealed, opaque envelopes. The principal investigator (PI), patients, and all other study personnel will remain concealed from the group assignments until the envelopes are opened.

   Due to the nature of the intervention, blinding of participants and intervention providers is not feasible. However, two outcome assessors will remain blinded to group allocation throughout the study to minimize detection bias.

   Outcome measures will be assessed at the same time points for both groups (baseline (T1), 2 weeks during intervention (T2), immediately after the intervention (T3), 4 weeks follow-up after the intervention (T4), and 8 weeks follow-up after the intervention (T5)), ensuring consistency in data collection across groups. All outcome evaluations will be performed by two assessors who are blinded to group allocation to minimize detection bias.

   After approval from the Institutional Review Board of Hanoi University of Public Health, the researcher will ask permission from the hospital to collect data. Data collection will take place across five time points, each aligned with a specific stage of the study process. During the initial visit, potential participants will be screened to determine eligibility based on inclusion and exclusion criteria. Prior to participation, all eligible individuals will be fully informed about the study procedures, potential risks and benefits, confidentiality measures, and their right to withdraw at any time without consequence. Only those who voluntarily agree to participate and sign the informed consent form will be enrolled in the study. Baseline outcome measures will then be collected using standardized instruments. In the second visit, participants will be randomized into 2 groups by opening the envelope in the order they are enrolled in the study. Participants in the intervention group will receive training on how to download, install, and operate the mobile application. At the end of the 2-week intervention period, participants will complete the same set of paper questionnaires to evaluate the short-term effects of the intervention. In the fourth visit, participants will complete paper-based outcome assessments to examine effects immediately after the intervention. The outcomes will be followed up at 4 and 8 weeks after the intervention.

   Patients will complete questionnaires by themselves or with assistance from two outcome assessors who will be blinded to group allocation. Both outcome assessors will receive a structured training program prior to initiating data collection to ensure standardized and unbiased assessment across study groups. Each questionnaire will be administered in a quiet and private area within the dialysis unit to ensure comfort and confidentiality. All completed paper forms will be reviewed on-site for completeness before being securely stored in locked cabinets accessible only to authorized study personnel. Data from the paper forms will later be entered into an Excel file by trained data entry staff.

   To promote participant retention and encourage full participation in the study, individuals will receive a total incentive of 300.000 dong (VND) (~12 USD) upon completion of all five data collection sessions. The incentive will be provided in cash after the final follow-up assessment. The study will be conducted from October 2025 to May 2026.
5. Statistical analysis The collected data will be analyzed using SPSS version 22.0 for Windows (IBM, Armonk, NY, USA). The general characteristics of each participant will be presented as frequency, percentage, and mean ± standard deviation (SD). Differences between the intervention and control groups at baseline will be analyzed using χ2-test, Fisher exact test, and the parametric tests (independent t-test, and one-way ANOVA) if the dependent variables meet assumptions of normality. If normality is not met, non-parametric tests (Mann-Whitney rank test, Kruskal-Wallis test) will be applied. Normality will be confirmed using skewness and kurtosis values, with acceptable ranges defines as skewness within ± 2 and kurtosis within ± 7, indicating a normal distribution (Byrne, 2010). If significant differences are found between groups at baseline, those variables will be considered as covariates in subsequent analyses. Both intention-to-treat and per-protocol analyses will be performed. Generalized Estimating Equations (GEE) analysis will be used to assess differences over time between groups and to adjust for potential covariates when necessary. In addition, a sensitivity analysis will be conducted to assess the impact of missing data, using multiple imputation with 10 sets of imputations.
6. Ethical approval The study protocol will be submitted to the Institutional Review Board of Hanoi University of Public Health, Hanoi, Vietnam for approval. The study will be conducted in accordance with the "Declaration of Helsinki". Participation in the study is entirely voluntary. An information sheet outlining the study's purpose, procedures, potential risks, and benefits is provided. Written informed consent will be obtained from all participants. Participants will be free to withdraw from the study at any time without any consequences.

ELIGIBILITY:
Inclusion Criteria: The patients are

* 18 years old or over
* are able to speak and understand Vietnamese,
* receive hemodialysis at least three times a week for three months or longer
* have a score equal to or greater than 4 on a numeric rating scale (NRS, 0-10)
* has a smartphone or tablet
* can provide written informed consent. Exclusion Criteria: The patients who have
* advanced cancer
* cognitive impairment
* chronic obstructive pulmonary disease
* severe edema
* have already used or plan to use acupressure or acupuncture in the following 3 months
* have soft tissue or vascular disease in their lower extremities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2026-03-15 (Estimated); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
Fatigue | Fatigue will be assessed at the same time points for both groups (baseline (T1), 2 weeks during intervention (T2), immediately after the intervention (T3), 4 weeks follow-up after the intervention (T4), and 8 weeks follow-up after the intervention (T5)).
  Fatigue will be measured by Post-dialysis fatigue (PDF) scale. This scale comprises 13 self-reported items rated on a five-point Likert scale, ranging from 1 (strongly agree) to 5 (not at all). The score will be reversed for analysis, and the total score is between 13 and 65, with higher scores indicating more severe fatigue.

SECONDARY OUTCOMES:
Pruritus | Pruritus will be assessed at the same time points for both groups (baseline (T1), 2 weeks during intervention (T2), immediately after the intervention (T3), 4 weeks follow-up after the intervention (T4), and 8 weeks follow-up after the intervention (T5))
  Pruritus will be measured by the 5-D Itch scale to evaluate the severity of skin itching conditions over the past 2 weeks based on five dimensions: duration, degree, direction, disability, and distribution. Itching at up to two sites receives a score of 1; three to five sites are assigned a score of 2; the score is 3 for six to ten sites; 11 to 13 sites are scored 4; and the highest score of 5 is given for 14 to 16 sites. The total scores range from 5 to 25. Higher scores indicate greater itch severity.
Sleep quality | Outcome will be assessed at the same time points for both groups (baseline (T1), 2 weeks during intervention (T2), immediately after the intervention (T3), 4 weeks follow-up after the intervention (T4), and 8 weeks follow-up after the intervention (T5)).
  Sleep quality will be measured by Pittsburgh Sleep Quality Index. The PSQI was developed by Buysse et al. (1989) consists of 7 components, 3 factors, and 19 subitems, and aims to evaluate a person's sleep quality within the last month, including seven components: (1) subjective sleep quality, (2) sleep latency, (3) sleep duration, (4) habitual sleep efficiency, (5) sleep disturbances, (6) use of sleeping medication and (7) daytime dysfunction. Component scores range from 0 (no difficulty) to 3 (severe difficulty). The total score ranges from 0 to 21, with higher values indicating poor sleep quality. A score of more than 5 indicated a person had poor quality sleep.

CONTACTS AND LOCATIONS:
Locations (1):
- Hoe Nhai General Hospital, Hanoi, Hong Ha, Vietnam

IPD SHARING:
Plan to Share IPD: No